CLINICAL TRIAL: NCT02440256
Title: The Expanded HIV Care in Opioid Substitution Treatment (EHOST) Stepped-wedge, Cluster-randomized Trial
Brief Title: Expanded HIV Care in Opioid Substitution Treatment (EHOST) Trial
Acronym: EHOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: BC Centre for Excellence in HIV/AIDS (Unknown)
Responsible Party: Principal Investigator, Bohdan Nosyk, Associate Professor, Faculty of Health Sciences, Health Economics; Endowed Chair in Health Economics HIV/AIDS, Simon Fraser University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: MOP313184
Record Dates: First submitted 2015-03-24; First posted 2015-05-12 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Opioid Use Disorder; HIV
Keywords: Cost-effectiveness; Opioid substitution treatment; Integrated care; HIV; HAART; Testing; Linkage to care; Treatment adherence
MeSH Terms: conditions — Opioid-Related Disorders; Treatment Adherence and Compliance | interventions — Opiate Substitution Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cluster 1 (Other): Cluster 1 is the first OST cluster (with an estimated 15-16 OST sites) to receive the 'Expanded HIV care in Opioid Substitution Treatment' intervention, to be administered during the sixth month of the trial. Cluster 1 will be a 'no intervention' arm in the first 6 months of the study, and will cross-over to an experimental arm for months 6-24.
  Interventions: Other: Expanded HIV care in Opioid Substitution Treatment
- Cluster 2 (Other): Cluster 2 is the second OST cluster (with an estimated 15-16 OST sites) to receive the 'Expanded HIV care in Opioid Substitution Treatment' intervention, to be administered during the twelfth month of the trial. Cluster 2 will be a 'no intervention' arm in the first 12 months of the study, and will cross-over to a experimental arm for month 12-24.
  Interventions: Other: Expanded HIV care in Opioid Substitution Treatment
- Cluster 3 (Other): Cluster 3 is the final OST cluster (with an estimated 15-16 OST sites) to receive the 'Expanded HIV care in Opioid Substitution Treatment' intervention, to be administered during the 18th month of the trial. As such, Cluster 3 will be a 'no intervention' arm in the first 18 months of the study, and will cross-over to an experimental arm for months 18-24.
  Interventions: Other: Expanded HIV care in Opioid Substitution Treatment

INTERVENTIONS:
Other: Expanded HIV care in Opioid Substitution Treatment — The EHOST intervention entails in-person presentations and consultation sessions with individual OST sites that will: (i) provide rationale for the study (ii) outline action items of the intervention; and (iii) describe guidelines around HIV testing and care. The EHOST intervention will be delivered at three distinct times: (i) at point of OST entry; (ii) following 7 days non-adherence; and (iii) at bi-annual intervals. The interventions are comprised of HIV test offers for individuals of unknown HIV status; offers of HIV-related care, including cluster of differentiation 4 (CD4), plasma viral load (pVL) and resistance tests, along with HAART initiation for those known to be HIV-positive, not on HAART; and regular monitoring for those known to be HIV positive, on HAART.

SUMMARY:
Opioid Substitution Treatment (OST) provides a critical opportunity for HIV testing and linkage to antiretroviral treatment. The EHOST study will evaluate a prescriber-focused intervention to increase HIV testing rates, and optimize antiretroviral treatment, re-engagement and retention outcomes among individuals engaged in OST. 46 OST sites in British Columbia will be randomly allocated into three clusters. Clusters will initiative the intervention at different time points, or steps, with every cluster receiving the intervention.

DETAILED DESCRIPTION:
The public health response to the HIV/AIDS epidemic has turned its focus on means of optimizing health care delivery, and re-engineering delivery systems to maximize case identification, as well as access and sustained engagement in antiretroviral treatment. Opioid Substitution Treatment (OST) provides a critical opportunity for HIV testing and linkage to antiretroviral treatment. The EHOST study is a cluster-randomized, stepped-wedge trial to evaluate a prescriber-focused intervention to increase HIV testing rates, and optimize antiretroviral treatment re-engagement and retention outcomes among individuals engaged in OST. The study will encompass all drug treatment clinics currently admitting patients for the treatment of opioid dependence across the province of British Columbia, which are thought to treat 90% of the OST caseload. The trial will be executed over a 24-month period, with groups of clinics receiving the intervention in 6-month intervals. Evaluation of the effectiveness of the proposed intervention will be conducted entirely through existing data collection mechanisms, and focuses on three primary outcomes: (i) the HIV testing rate among those not known to be HIV positive; (ii) the rate of Highly Active Antiretroviral (HAART) initiation among those not on HAART; and (iii) the rate of HAART continuation among those on HAART. Despite the randomized delivery of the intervention, a difference-in-differences analytical framework will be applied to adjust for potential residual heterogeneity in patient case mix, volume, and quality of care across OST clinics. Facilitated by established collaborations between key stakeholders across the province, we hypothesize that the EHOST intervention will optimize HIV testing and care within this marginalized and hard-to-reach population.

ELIGIBILITY:
Inclusion Criteria:

* Drug treatment clinic currently admitting patients for the treatment of opioid dependence across the province of British Columbia

Exclusion Criteria:

* Private office-based setting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The HIV testing rate among those not known to be HIV positive | 24 months
The rate of Highly Active Antiretroviral (HAART) initiation among those not on HAART | 24 months
The rate of HAART adherence among those on HAART | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan Nosyk, PhD, Principal Investigator — Simon Fraser University